CLINICAL TRIAL: NCT00278941
Title: A Multi-Centre, Double-Blind, Randomised-Withdrawal, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (SEROQUEL SR™) As Monotherapy in the Maintenance Treatment of Patients With Major Depressive Disorder
Brief Title: Quetiapine Fumarate as Monotherapy in the Maintenance Treatment of Patients With Major Depressive Disorder
Acronym: AMETHYST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00005; Amethyst
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: Seroquel SR™; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: Quetiapine Fumarate Sustained Release

SUMMARY:
The purpose of this study is to determine safety & efficacy of SEROQUEL SR™ in the treatment of major depressive disorder compared to placebo & to evaluate quality of sleep, overall quality of life, and effect, if any, on anxiety and satisfaction PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis according to the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision) meeting criteria 296.2x Major Depressive Disorder,
* Single Episode, or 296.3x Major Depressive Disorder,

Exclusion Criteria:

* Patients with a DSM-IV Axis I disorder other than MDD w/in 6 months of enrollment,
* Patients with a diagnosis of DSM-IV Axis II disorder which has a major impact on the patients current psychiatric status.
* Patients whose current episode of depression>12 months or <4 weeks from enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2005-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of quetiapine SR compared to placebo in increasing time from randomisation to a depressed event in patients with Major Depressive Disorder (MDD)

SECONDARY OUTCOMES:
Evaluate quetiapine SR compared to placebo on health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (168):
- United States (144):
  - Research Site, Birmingham, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Costa Mesa, California
  - Research Site, El Centro, California
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Pasadena, California
  - Research Site, Pico Rivera, California
  - Research Site, Redlands, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Stanford, California
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Vista, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Pueblo, Colorado
  - Research Site, Cromwell, Connecticut
  - Research Site, Farmington, Connecticut
  - Research Site, Middletown, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, North Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Saint Petersberg, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Stuart, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Sandy Springs, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Granite City, Illinois
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Libertyville, Illinois
  - Research Site, Northfield, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Terre Haute, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Glen Burnie, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Cambridge, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Clinton Twp, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Portage, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Flowood, Mississippi
  - Research Site, Ridgeland, Mississippi
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Kenilworth, New Jersey
  - Research Site, Princeton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Cedarhurst, New York
  - Research Site, Mount Kisco, New York
  - Research Site, New York, New York
  - Research Site, Olean, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Avon Lake, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Chagrin Falls, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Coatesville, Pennsylvania
  - Research Site, Havertown, Pennsylvania
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Media, Pennsylvania
  - Research Site, Moon Township, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, DeSoto, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Houston, Texas
  - Research Site, Lake Jackson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Midvale, Utah
  - Research Site, Woodstock, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Vratsa, Bulgaria
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Miramichi, New Brunswick
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Research Site, Rio Predia, Puerto Rico
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Piteşti
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (4):
  - Research Site, Piešťany
  - Research Site, Prešov
  - Research Site, Sereď
  - Research Site, Trenčín
- United Kingdom (3):
  - Research Site, Ayrshire
  - Research Site, Glasgow
  - Research Site, Reading

REFERENCES:
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS. The role of extended-release quetiapine fumarate monotherapy in the treatment of patients with major depressive disorder. Expert Rev Neurother. 2013 Nov;13(11):1161-82. doi: 10.1586/14737175.2013.846520. PMID 24175720